CLINICAL TRIAL: NCT05231759
Title: Efficacy of Navigable Percutaneous Plasma Disc Decompression Device (L'DISQ) in Patients With Severe Lumbar Disc Herniation
Acronym: L'DISQ
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K2021-2858-001
Record Dates: First submitted 2022-01-21; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Lumbar Disc Herniation
Keywords: Low Back Pain; Percutaneous Decompression; Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Navigable Percutaneous Plasma Disc Decompression (L'DISQ): The L'DISQ (U&I Co., Uijeongbu, Korea) is one of the minimally invasive disc decompression procedures which was introduced in 2011. The L'DISQ uses a navigable tip and flexible handle allowing resection of the posterolateral or posterior median disc tissue without thermal damage.
  Interventions: Device: L'DISQ

INTERVENTIONS:
Device: L'DISQ

SUMMARY:
This study aims to assess the clinical outcome of percutaneous disc decompression using the L'DISQ in patients with severe lumbar disc herniation (LDH).

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most leading cause of chronic pain worldwide and 70-85% of adults have experienced LBP during their lifetime. The one of most common symptom of lumbar disc herniation (LDH) is sciatica, affecting about 1-5% of people worldwide. Almost two thirds of patients suffer from continuous pain even after 12 months of the first episode of LBP. Moreover, such persistent pain reduces the patient's quality of life and increases the social and economic burden due to increased hospital stay and surgical treatment. Traditionally, the primary treatment of LDH is non-surgical treatment including pain medication, rehabilitation exercise, and spinal injection, and about 70% of the patients show improvement of pain within 4 weeks. Surgical treatment is considered if there are neurological symptoms such as bladder dysfunction or progressive muscle weakness, or if symptoms persist for more than 6 weeks despite conservative treatment.

The patients with LDH usually experience sudden onset of LBP with radiating pain to lower extremity. Sensory symptoms such as focal paresis or motor weakness of specific myotome can also occur in the LDH patients. The symptoms and area of pain can vary due to the herniation level and severity. Michigan State University (MSU) classification was often used to evaluate and select for surgical treatment of LDH patients. In this classification, the herniated disc is evaluated using T2 axial magnetic resonance imaging (MRI) scan and classified by its size and location. The size of disc herniation is classified into 1 (*<50% of the distance to the intra-facet line), 2 (intra-facet line>*≥50% of the distance to the intra-facet line), or 3 (beyond intra-facet line). Then the position is classified in to A (central), B (lateral), or C (far lateral). The disc herniations size 3 (beyond intra-facet line) and zone B (lateral) or C (far lateral) are known to have greater impact on nerve compression, which tend to cause worse sciatica and neurologic symptoms and require surgical treatment. Moreover, the patients with larger lumbar disc herniation areas tend to show better outcomes with surgical treatment than conservative treatments and high-grade spinal canal stenosis patients had higher need for surgical treatment.

Over the past few years, various minimally invasive disc decompression procedures, were developed and used in LDH patients. These minimally invasive disc decompression techniques include intradiscal electrothermal therapy, radiofrequency annuloplasy, percutaneous disc decompression, nucleoplasty, and percutaneous laser disc decompression, which caused less damage to spinal structures and reduced tissue destructions than conventional surgical treatments. In particular, nucleoplasty was proven as effective as open discectomy in the treatment of single level lumbar disc herniation. The L'DISQ (U&I Co., Uijeongbu, Korea) is one of the safe and effective minimally invasive disc decompression procedures which introduced in 2011. In contrast to most percutaneous nucleotomy procedures that used rigid tip, the L'DISQ used a navigable tip and flexible handle allowing resection of the posterolateral or posterior median disc tissue without thermal damage.

The L'DISQ can be mainly performed in patients with less severe LDH while surgical treatment was mainly indicated in patients with severe LDH with neurologic symptoms. However, surgical treatment such as lumbar discectomy or spinal fusion increase hospitalization time and may increase financial burden of patients. And spinal fusion surgery might lead to delayed complications such as back muscle weakness or adjacent segment disease. Moreover, patients with severe LDH might refuse or not be able to perform surgery due to medical, financial, or other personal reasons. Recently, studies on the efficacy of L'DISQ or plasma decompression in disc patients are being conducted, and shows similar outcome when compared to surgical treatment in mild to moderate disc herniation patients. However, no studies have been conducted on the efficacy of L'DISQ in patients with severe LDH requiring surgical treatment. Purpose of this study is to report the efficacy of the L'DISQ procedure in patients with severe LDH corresponding to MSU classification 3.

ELIGIBILITY:
Inclusion Criteria:

1. single-level LDH of MSU classification of grade 3 and refusal of spine surgery
2. LBP or lower extremity pain symptoms that persisted for 3 months or more
3. unresponsiveness to sufficient conservative treatments, including oral analgesics, physical modalities, or spinal injections (such as selective nerve root blocks)
4. limited activities of daily living due to pain.

Exclusion Criteria:

1. patients lost during the 1-year follow-up
2. evidence of peripheral neuropathy on electromyography, which might cause lower extremity pain
3. evidence of vertebral fracture in the X-ray analysis
4. history of tumor or myelopathy
5. history of spinal surgery
6. history of coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have visited the spine center of Korea University Anam Hospital and received the L'DISQ procedure between March 01, 2009 and February 28, 2019
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Change from baseline data, evaluated during the hospitalization prior to the L'DISQ procedure, to 4, 12, 24, and 48 weeks after the procedure.
  VAS (Visual Analogue Scale) is a measuring tool that can quickly and easily measure the level of pain through the patient's expression or attitude.

SECONDARY OUTCOMES:
Straight Leg Raise Test (SLRT) | Change from baseline data, evaluated during the hospitalization prior to the L'DISQ procedure, to 4, 12, 24, and 48 weeks after the procedure
  The SLRT is a test that measures the initial angle at which the patient complains of lower extremity radiating pain during the passive hip flexion with knee extended in supine position. Normal people show hip flexion angle of 80 to 90 degrees, but the hip flexion angle at the initiationg of pain is reduced in LDH patients due to nerve irritation at the level of disc prolapse
Roland-Morris Disability Questionnaire (RMDQ) | Change from baseline data, evaluated during the hospitalization prior to the L'DISQ procedure, to 4, 12, 24, and 48 weeks after the procedure
  The RMDQ is used to evaluate physical disability caused by low back pain and its score range from 0 to 24. The higher score means greater level of disability
Oswestry Disability Index (ODI) | Change from baseline data, evaluated during the hospitalization prior to the L'DISQ procedure, to 4, 12, 24, and 48 weeks after the procedure
  The ODI is used to assess chronic low back pain symptoms and is consisted of 10 questions. The ODI score can result from 0 to 100% and higher score also means greater level of disabilities.
Physical Component Score (PCS) of Short Form-36 version 2 (SF-36v2) | Change from baseline data, evaluated during the hospitalization prior to the L'DISQ procedure, to 4, 12, 24, and 48 weeks after the procedure
  The PCS is component of SF-36v2. The SF-36v2 is a short-form survey for evaluating health status including physical and mental factors. The PCS shows summary of physical component. It can be scored from 0 to 100 and higher scores indicates better health status.
Bodily Pain Score (BPS) of Short Form-36 version 2 (SF-36v2) | Change from baseline data, evaluated during the hospitalization prior to the L'DISQ procedure, to 4, 12, 24, and 48 weeks after the procedure
  The BPS is component of SF-36v2. The SF-36v2 is a short-form survey for evaluating health status including physical and mental factors. The BPS shows summary of bodily pain component. It can be scored from 0 to 100 and higher scores indicates better health status.